CLINICAL TRIAL: NCT03321370
Title: Cortical Spreading Depolarization After Severe Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Principal Investigator, Samuel Cramer, Neurosurgery Attending Physician, Hennepin County Medical Center, Minneapolis
Other Study IDs: HSR 17-4400
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Continuous electrocorticography post severe traumatic brain injury requiring neurosurgical intervention — Continuous electrocorticography via subdural electrode strips for 1 to 3 weeks in the neuro intensive care unit following traumatic brain injury

SUMMARY:
Preliminary evaluation of electrodes placed on the brain for recording brain activity and novel algorithms to determine cortical spreading depolarization foci of origination following severe traumatic brain injury requiring neurosurgical intervention.

DETAILED DESCRIPTION:
The goal of this study is to improve our understanding of cortical spreading depolarizations (CSDs) as a mechanism of secondary injury in severe traumatic brain injury (TBI). The primary obstacles to advancing treatment of TBI are its heterogeneity in terms of cause, severity, pathophysiology and the paucity of therapeutic targets. At the current time, there is no intervention to reverse or restore the function of brain tissue damaged or lost during the initial traumatic insult; therefore the therapeutic focus is centered on minimizing secondary insults that result in expansion of the initial brain injury.

The past several years have witnessed significant advancement in the understanding of potential mechanisms of secondary injury after severe TBI. This is important work as secondary injury after severe TBI is thought to significantly increase the severity of the initial injury and this type of injury is thought to be open to interventions to attenuate the subsequent injury severity. Among the putative mechanisms of secondary injury after severe TBI, it was recently demonstrated that there is a relationship between CSD events and worse outcomes after severe TBI. Therefore, a more thorough understanding of the factors that influence the initiation and frequency of CSDs after TBI is warranted in order to develop therapeutic strategies to reduce or block these events from occurring.

In young people, TBI is the leading cause of morbidity and mortality in developed countries. TBI is a frequent sequelae of accidental injury in the USA with approximately 2.5 million people affected per year, approximately 10% of whom requiring extended hospitalization, often in an intensive care unit. Around 275,000 (15.1%) of hospital admissions and 52,000 deaths in the USA each year are due to TBI. Those that survive the initial insult invariably face prolonged stays in a neurologic intensive care unit (ICU), possible neurosurgical intervention, and prolonged period of post-acute supportive care. In the US, it is estimated that 5.3 million individuals are living with long-term disability as a result of TBI.

Given the complexity and duration of medical care that accompanies severe TBI, it follows that the cost of care associated with TBI are immense. It is estimated that total hospital charges for TBI-related admissions in 2010 were $21.4 billion. Beyond hospital charges, it is estimated that TBI costs the US economy $76.5 billion annually with the costs for disability and lost productivity outweighing those of acute medical care and rehabilitation.

Since their first description in 1944, spreading depolarizations (SDs) were subsequently demonstrated in numerous animal studies as a mechanism of secondary brain injury after ischemic stroke, subarachnoid hemorrhage (SAH), and traumatic brain injury. SDs have also been demonstrated to occur in the cerebral grey matter of the human brain in patients after acute brain injuries such as TBI, SAH, and ischemic stroke. To date, electrocorticography (ECoG) monitoring of over 500 patients after TBI has shown that SDs occur in 55-90% of individuals for days to weeks after the initial injury. These studies have demonstrated an initial peak in SD frequency at 1-2 days post-TBI and a second peak at 6-7 days. Furthermore, SDs are associated with worse outcomes after TBI.

SDs which consist of massive waves that depolarize neurons and astrocytes and disrupt local cortical function for minutes to hours, were first demonstrated to occur in severe TBI patients via ECoG recordings obtained from single subdural electrode strips. In these studies, severe TBI patients who underwent neurosurgical intervention for decompression and/or hematoma evacuation had a single linear subdural electrode strips (six electrodes with 10 mm spacing between electrodes) placed near the injury epicenter which allowed continuous ECoG recordings to be obtained for up to 7 days after the initial injury. The above studies, and several subsequent investigations, were important steps to demonstrate that (1) the SD phenomena, which was first described in animal studies, occurs in patients after TBI and (2) SDs are associated with worse outcome after TBI.

Despite the advances that have been made, previous studies discontinued ECoG recordings after a maximum of 7 days. A 7 day recording period is, however, likely inadequate to accurately characterize the total burden of SDs following TBI as previous work demonstrates an early peak period of SDs around 0-2 days post-TBI followed by a relative quiescent period and then a second peak of increased SD frequency around 7 days post-TBI. Therefore, a longer recordings period will provide a better understanding of the natural history of SDs following TBI and allow a more accurate understanding of the physiologic and pathophysiologic factors that influence initiation of these pathologic events.

All prior ECoG recordings of SDs has relied on subdural electrode strips consisting of a linear array of electrodes placed over the cerebral cortex near contused brain tissue. This recordings strategy is adequate to capture SD events, however, it affords the ability to monitor a small area of the cortical surface. The small monitoring area imposed several limitations on previous studies. First, CSDs are captured within a limited distance of each recording electrode contact. CSDs that occur beyond the monitoring region are not recorded and, therefore, prior studies likely underestimate the true frequency of SD events after TBI. Second, the linear configuration of subdural strips does not provide adequate spatial information regarding the CSD waves to determine the origin or direction of propagation. Improved spatial resolution of the ECoG recordings in conjunction with appropriate analytic techniques will allow determination of the direction of SD wave propagation and possibly the identification of pathologic foci where SDs originate. Identification of where SDs originate will afford the ability to correlate these locations with imaging to determine the structural characteristics and pathology that give rise to this pathological phenomenon.

The overall goal of this study is to preliminarily evaluate an improved recording strategy and analytical techniques to better define SD events and structural abnormalities in the severely injured brain that produce these CSD events in severe TBI. In order to achieve this goal, this study will utilize 4 subdural electrode strips arranged to produce a 4x4 grid of electrode contacts for the recording of ECoG activity in conjunction with simultaneous acquisition of several other physiological measures in TBI patients requiring neurosurgical intervention.

The findings of this study could provide a key advancement in the means to both monitor CSD events after TBI and identify the specific types of pathology that give rise to these events. This would be an important next step in the development of new interventions to reduce or eliminate the frequency of SDs in TBI patients and thus the degree of secondary brain injury that leads to greater morbidity and mortality after severe brain injury.

Despite advances that have been made in the care of patients after severe brain injury, TBI continues to confer a very high morbidity and mortality. The development of effective treatments to minimize the morbidity and mortality following TBI has been hindered due to a fundamental lack of understanding of the factors that contribute to secondary injury after the initial inciting traumatic event. By better understanding mechanisms of secondary brain injury after TBI, such as CSD, as well as methods for monitoring for pathologic events, there will be more opportunities to develop new treatments. This is a preliminary study with the goal of better characterizing CSD following severe TBI.

Subdural electrodes have been used extensively to record ECoG activity following TBI and other forms of brain injury. Despite requiring an invasive form of recording, ECoG activity remains the only established means to monitor CSD events. Invasive neuromonitoring via subdural electrodes was first demonstrated in the 1930s and continues to be a commonly performed neurosurgical procedure for epilepsy monitoring. A recent retrospective review found an overall complication rate of approximately 9.1% with 0.6% of patients experiencing permanent neurological deficits following subdural electrode placement.19 Furthermore, there has not been a single infection associated with subdural electrode placement at the University of Minnesota Medical Center. In addition to allowing detection of CSD events, subdural electrodes will allow the identification of subclinical seizures, and, therefore may provide a clinical benefit to the patients who undergo subdural electrode recording.

Subjects enrolled in this study will be selected from patients requiring neurosurgical intervention in the form of craniectomy or craniotomy and, therefore, will not be exposed to an invasive procedure solely for the placement of subdural recording electrodes. During the standard craniectomy/craniotomy procedure, the dura is opened to expose allowing the placement of the subdural recording strips with minimal modification to the standard surgical procedure. After the subdural strips are placed, the leads will be tunneled away from the brain so that they exit away from the brain, minimizing infection risk. This approach has the added benefit that when the study period is over, the tunneled leads can be removed at the bedside.

In addition to ECoG recordings, other forms of invasive neuromonitoring, including Licox bolt (Integra Life Sciences, Plainsboro, New Jersey) for measurement of ICP, brain tissue oxygenation and temperature, as well as external ventricular drain (EVD) will be placed as part of the current standard of care treatment for severe TBI.

The study period will be as long as invasive neuromonitoring is clinically indicated following severe TBI. As outlined in the background section, previous investigations of CSD have ended after a 7-day recording period. The shorter recording period has likely hindered a full understanding of the natural history of CSDs following severe TBI and therefore a full understanding of the pathophysiological factors that produce these events. There will be minimal additional risk to extending the recording period to the full period of clinically indicated invasive neuromonitoring as subdural recording is routinely performed at the University of Minnesota for epilepsy monitoring for 4-6 weeks without a documented serious complication.

Hennepin County Medical Center (HCMC) is a regional level 1 trauma center that serves the upper midwest and is one of the training sites for the University of Minnesota Neurosurgery Residency Program. As a large regional trauma center, there has historically been a large volume of severe TBI patients requiring neurosurgical intervention in the form of craniectomy or craniotomy with subsequent prolonged invasive neuromonitoring necessary as part of the clinical standard of care. The study population will be drawn from all trauma patients who present to the HCMC Emergency Department, trauma bay or as direct transfer to neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient recommended to undergo craniectomy or craniotomy for the treatment of acute TBI

Exclusion Criteria:

* Wound determined to be contaminated
* Decompression is performed only in the posterior fossa
* Known systemic infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the population of severe TBI patients clinically judged to require neurosurgical intervention who present through the emergency department or upon direct transfer to the neurosurgery service at Hennepin County Medical Center. The target sample size for this preliminary study is 10 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Determination of foci that give rise to cortical spreading depolarizations | 2 years

SECONDARY OUTCOMES:
Determine the relationship between cortical spreading depolarization foci of origination and structural pathology demonstrated on brain imaging (CT and MRI). | 2 years

OTHER OUTCOMES:
Determine the association (if any) between cortical spreading depolarization foci of origination and cortical spreading depolarization frequency with relevant physiological data. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel W Cramer, MD, PhD, Principal Investigator — University of Minnesota Neurosurgery Department; Division of Neurosurgery, Department of Surgery, Hennepin County Medical Center
Locations (1):
- Hennepn Healthcare, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, individual participant data that underlie the results reported in study publications (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 36 months following article publication.
Access Criteria: To investigators who provide a methodologically sound proposal whose proposed use of data has been approved by an independent review committee for the proposed purpose. Data requests should be directed to the corresponding author of the publication that forms the basis for the data requests. Investigators will have to sign a data use agreement in order to gain access to the data.

REFERENCES:
- [Background] Dreier JP, Fabricius M, Ayata C, Sakowitz OW, Shuttleworth CW, Dohmen C, Graf R, Vajkoczy P, Helbok R, Suzuki M, Schiefecker AJ, Major S, Winkler MK, Kang EJ, Milakara D, Oliveira-Ferreira AI, Reiffurth C, Revankar GS, Sugimoto K, Dengler NF, Hecht N, Foreman B, Feyen B, Kondziella D, Friberg CK, Piilgaard H, Rosenthal ES, Westover MB, Maslarova A, Santos E, Hertle D, Sanchez-Porras R, Jewell SL, Balanca B, Platz J, Hinzman JM, Luckl J, Schoknecht K, Scholl M, Drenckhahn C, Feuerstein D, Eriksen N, Horst V, Bretz JS, Jahnke P, Scheel M, Bohner G, Rostrup E, Pakkenberg B, Heinemann U, Claassen J, Carlson AP, Kowoll CM, Lublinsky S, Chassidim Y, Shelef I, Friedman A, Brinker G, Reiner M, Kirov SA, Andrew RD, Farkas E, Guresir E, Vatter H, Chung LS, Brennan KC, Lieutaud T, Marinesco S, Maas AI, Sahuquillo J, Dahlem MA, Richter F, Herreras O, Boutelle MG, Okonkwo DO, Bullock MR, Witte OW, Martus P, van den Maagdenberg AM, Ferrari MD, Dijkhuizen RM, Shutter LA, Andaluz N, Schulte AP, MacVicar B, Watanabe T, Woitzik J, Lauritzen M, Strong AJ, Hartings JA. Recording, analysis, and interpretation of spreading depolarizations in neurointensive care: Review and recommendations of the COSBID research group. J Cereb Blood Flow Metab. 2017 May;37(5):1595-1625. doi: 10.1177/0271678X16654496. Epub 2016 Jan 1. PMID 27317657
- [Background] Dreier JP, Woitzik J, Fabricius M, Bhatia R, Major S, Drenckhahn C, Lehmann TN, Sarrafzadeh A, Willumsen L, Hartings JA, Sakowitz OW, Seemann JH, Thieme A, Lauritzen M, Strong AJ. Delayed ischaemic neurological deficits after subarachnoid haemorrhage are associated with clusters of spreading depolarizations. Brain. 2006 Dec;129(Pt 12):3224-37. doi: 10.1093/brain/awl297. Epub 2006 Oct 25. PMID 17067993
- [Background] Drenckhahn C, Windler C, Major S, Kang EJ, Scheel M, Vajkoczy P, Hartings JA, Woitzik J, Dreier JP; COSBID study group. Complications in Aneurysmal Subarachnoid Hemorrhage Patients With and Without Subdural Electrode Strip for Electrocorticography. J Clin Neurophysiol. 2016 Jun;33(3):250-9. doi: 10.1097/WNP.0000000000000274. PMID 27258449
- [Background] Fabricius M, Fuhr S, Bhatia R, Boutelle M, Hashemi P, Strong AJ, Lauritzen M. Cortical spreading depression and peri-infarct depolarization in acutely injured human cerebral cortex. Brain. 2006 Mar;129(Pt 3):778-90. doi: 10.1093/brain/awh716. Epub 2005 Dec 19. PMID 16364954
- [Background] Hartings JA, Bullock MR, Okonkwo DO, Murray LS, Murray GD, Fabricius M, Maas AI, Woitzik J, Sakowitz O, Mathern B, Roozenbeek B, Lingsma H, Dreier JP, Puccio AM, Shutter LA, Pahl C, Strong AJ; Co-Operative Study on Brain Injury Depolarisations. Spreading depolarisations and outcome after traumatic brain injury: a prospective observational study. Lancet Neurol. 2011 Dec;10(12):1058-64. doi: 10.1016/S1474-4422(11)70243-5. Epub 2011 Nov 3. PMID 22056157
- [Background] Hartings JA, Li C, Hinzman JM, Shuttleworth CW, Ernst GL, Dreier JP, Wilson JA, Andaluz N, Foreman B, Carlson AP. Direct current electrocorticography for clinical neuromonitoring of spreading depolarizations. J Cereb Blood Flow Metab. 2017 May;37(5):1857-1870. doi: 10.1177/0271678X16653135. Epub 2016 Jan 1. PMID 27286981
- [Background] Hartings JA, Shuttleworth CW, Kirov SA, Ayata C, Hinzman JM, Foreman B, Andrew RD, Boutelle MG, Brennan KC, Carlson AP, Dahlem MA, Drenckhahn C, Dohmen C, Fabricius M, Farkas E, Feuerstein D, Graf R, Helbok R, Lauritzen M, Major S, Oliveira-Ferreira AI, Richter F, Rosenthal ES, Sakowitz OW, Sanchez-Porras R, Santos E, Scholl M, Strong AJ, Urbach A, Westover MB, Winkler MK, Witte OW, Woitzik J, Dreier JP. The continuum of spreading depolarizations in acute cortical lesion development: Examining Leao's legacy. J Cereb Blood Flow Metab. 2017 May;37(5):1571-1594. doi: 10.1177/0271678X16654495. Epub 2016 Jan 1. PMID 27328690
- [Background] Hartings JA, Strong AJ, Fabricius M, Manning A, Bhatia R, Dreier JP, Mazzeo AT, Tortella FC, Bullock MR; Co-Operative Study of Brain Injury Depolarizations. Spreading depolarizations and late secondary insults after traumatic brain injury. J Neurotrauma. 2009 Nov;26(11):1857-66. doi: 10.1089/neu.2009.0961. PMID 19508156
- [Background] Hartings JA, Watanabe T, Bullock MR, Okonkwo DO, Fabricius M, Woitzik J, Dreier JP, Puccio A, Shutter LA, Pahl C, Strong AJ; Co-Operative Study on Brain Injury Depolarizations. Spreading depolarizations have prolonged direct current shifts and are associated with poor outcome in brain trauma. Brain. 2011 May;134(Pt 5):1529-40. doi: 10.1093/brain/awr048. Epub 2011 Apr 7. PMID 21478187
- [Background] Hinzman JM, Andaluz N, Shutter LA, Okonkwo DO, Pahl C, Strong AJ, Dreier JP, Hartings JA. Inverse neurovascular coupling to cortical spreading depolarizations in severe brain trauma. Brain. 2014 Nov;137(Pt 11):2960-72. doi: 10.1093/brain/awu241. Epub 2014 Aug 24. PMID 25154387
- [Background] Hinzman JM, Wilson JA, Mazzeo AT, Bullock MR, Hartings JA. Excitotoxicity and Metabolic Crisis Are Associated with Spreading Depolarizations in Severe Traumatic Brain Injury Patients. J Neurotrauma. 2016 Oct 1;33(19):1775-1783. doi: 10.1089/neu.2015.4226. Epub 2016 Mar 18. PMID 26586606
- [Background] Jeffcote T, Hinzman JM, Jewell SL, Learney RM, Pahl C, Tolias C, Walsh DC, Hocker S, Zakrzewska A, Fabricius ME, Strong AJ, Hartings JA, Boutelle MG. Detection of spreading depolarization with intraparenchymal electrodes in the injured human brain. Neurocrit Care. 2014 Feb;20(1):21-31. doi: 10.1007/s12028-013-9938-7. PMID 24343564
- [Background] Maas AI, Stocchetti N, Bullock R. Moderate and severe traumatic brain injury in adults. Lancet Neurol. 2008 Aug;7(8):728-41. doi: 10.1016/S1474-4422(08)70164-9. PMID 18635021
- [Background] Marin JR, Weaver MD, Mannix RC. Burden of USA hospital charges for traumatic brain injury. Brain Inj. 2017;31(1):24-31. doi: 10.1080/02699052.2016.1217351. Epub 2016 Nov 10. PMID 27830939
- [Background] Marin JR, Weaver MD, Yealy DM, Mannix RC. Trends in visits for traumatic brain injury to emergency departments in the United States. JAMA. 2014 May 14;311(18):1917-9. doi: 10.1001/jama.2014.3979. No abstract available. PMID 24825648
- [Background] Schmidt RF, Wu C, Lang MJ, Soni P, Williams KA Jr, Boorman DW, Evans JJ, Sperling MR, Sharan AD. Complications of subdural and depth electrodes in 269 patients undergoing 317 procedures for invasive monitoring in epilepsy. Epilepsia. 2016 Oct;57(10):1697-1708. doi: 10.1111/epi.13503. Epub 2016 Aug 23. PMID 27549686
- [Background] Strong AJ, Fabricius M, Boutelle MG, Hibbins SJ, Hopwood SE, Jones R, Parkin MC, Lauritzen M. Spreading and synchronous depressions of cortical activity in acutely injured human brain. Stroke. 2002 Dec;33(12):2738-43. doi: 10.1161/01.str.0000043073.69602.09. PMID 12468763
- [Background] Waxweiler RJ, Thurman D, Sniezek J, Sosin D, O'Neil J. Monitoring the impact of traumatic brain injury: a review and update. J Neurotrauma. 1995 Aug;12(4):509-16. doi: 10.1089/neu.1995.12.509. No abstract available. PMID 8683602
- [Derived] Cramer SW, Pino IP, Naik A, Carlson D, Park MC, Darrow DP. Mapping spreading depolarisations after traumatic brain injury: a pilot clinical study protocol. BMJ Open. 2022 Jul 13;12(7):e061663. doi: 10.1136/bmjopen-2022-061663. PMID 35831043